CLINICAL TRIAL: NCT05937802
Title: Exploratory Trial of Forza™️, a Novel Nutraceutical From Actinidia Deliciosa Plants Bioengineered to Bio-encapsulate the Osmotin Plant Protein as Adjuvant for the Treatment of Progressive Multiple Sclerosis
Brief Title: Osmotin Plant Protein for Progressive Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Collaborators: Italian Multiple Sclerosis Foundation (Other); S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Matilde Inglese, Clinical Professor, Principal Investigator, Ospedale Policlinico San Martino
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12042
Record Dates: First submitted 2023-05-22; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Osmotin
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osmotin (Experimental): Administration of a nutraceutical supplement provided in capsules, that consists of lyophilised and pulverised kiwi leaves from bioengineered kiwi (Actinidia Deliciosa) plants overexpressing the tobacco protein Osmotin.
  Interventions: Dietary Supplement: Osmotin

INTERVENTIONS:
Dietary Supplement: Osmotin — Oral administration for 6 months of 7 capsules per day (4 in the morning and 3 in the evening) for a daily dosage of 5 grams.
  Other Names: FORZA™️

SUMMARY:
The aim of this study is to explore the anti-inflammatory and neuroprotective effects of a novel nutraceutical product (commercial name Forza™️), consisting of the plant osmotin protein, in patients with progressive multiple sclerosis (PMS). The potential effect on brain metabolism and microstructure will be evaluated by magnetic resonance imaging (MRI) performed six months before starting treatment, at baseline, and after one and six months of treatment. At the same timepoints, electrophysiology, neurofilaments (NfL) quantification, optical coherence tomography (OCT) and clinical assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Diagnosis of progressive multiple sclerosis (PMS)
* Expanded Disability Status Scale EDSS ≤ 6.5

Exclusion Criteria:

* Contraindications to MRI
* Pregnancy
* HIV positivity
* Severe renal, hepatic, oncological, hematological and psychiatric diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-01-02 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-related adverse events after 1 month of therapy. | 1 month (after 1 month of treatment).
Incidence and severity of treatment-related adverse events after 6 months of therapy. | 6 months (after 6 months of treatment).

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS). | 12 months (6 month before starting treatment, at baseline and both after one month and six months of treatment)
  The EDSS score ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Change in Timed 25 Foot Walk (T25FW). | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Quantitative mobility and leg function performance test based on a timed 25-walk. T25FW improvement is ≥15% decrease in time from first record and worsening is ≥15% increase in time from first record.
Change in 12-item Multiple Sclerosis Walking Scale (MSWS12). | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Self-reported measure of the impact of Multiple Sclerosis on the individual's walking ability. The scoring provides 1-5 for each of the 12 items, with 1 meaning no limitations and 5 meaning extreme limitation, for a maximum total score of 60. Then, this total score is transformed to a scale with a range from 0 to 100. Higher scores indicate a greater impact on walking than lower scores.
Change in Nine-Hole Peg Test (9HPT). | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Quantitative measure of upper extremity (arm and hand) function. 9HPT improvement is ≥15% decrease in time from first record and worsening is ≥15% increase in time from first record.
Change in Montreal Cognitive Assessment (MOCA). | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Test to assesses different cognitive dimensions including attention and concentration, executive functions, memory, language, visuospatial skills, abstract thinking, calculation, and orientation. The lowest score that can be obtained from the scale is 0, and the highest score is 30. Higher scores indicate a better cognitive levels.
Change in Symbol Digit Modalities Test (SDMT). | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Test to assess cognitive processes including memory, lexical access speed and information processing speed. The score is the number of correct answers in 90 seconds. The total score ranged from 0 to 110. Higher values represent better outcome.
Change in patient self-evaluation of depression and anxiety recorded with Hospital Anxiety Depression Scale (HADS). | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Hospital Anxiety Depression Scale (HADS) is a 14 item questionnaire which consists two sub-scale evaluating anxiety (HADS-A) and depression (HADS-D).
  HADS-A sub-scale has seven items and each item is scored on a scale of 0 to 3. Total sub-scale score ranged from 0 to 21. Higher score mean a worse outcome.
  HADS-D sub-scale has seven items and each item is scored on a scale of 0 to 3. Total score ranged from 0 to 21. Higher scores reflects more severe depression.
Change in bladder domain function recorded with Overactive Bladder (OAB) questionnaire. | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Self-reported questionnaire to quantify Overactive Bladder symptoms including urgency, urination, frequent urination and feeling of urine at night and waking up. The scale consists of 8 items and answers are scored on a 6-level Likert scale. A maximum score of 40 can be obtained from the scale, and a score below 8 eliminates overactive bladder.
The impact of Forza™️ on neurophysiology in PMS. | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Motor evoked potentials (MEPs), somatosensory evoked potentials (SEPs), visual evoked potentials (VEPs) will be measured and compared pre and post treatment.
The impact of Forza™️ on retinal atrophy in PMS. | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Optical Coherence Tomography (OCT) will be measured and compared pre and post treatment to assess the retinal thickness.
Change in serum neurofilament Light Chain (NfL) levels to verify the neuroprotective action of Forza™️ in PMS. | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
Change in brain metabolism as concentration of glutamate, N-acetylaspartate, creatine and choline. | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Proton magnetic resonance spectroscopy (1H-MRI) will be performed to quantify brain glutamate, N-acetylaspartate, creatine and choline.
Change in brain microstructure. | 12 months (6 months before starting treatment, at baseline and both after one month and six months of treatment)
  Brain magnetic resonance imaging (MRI) will be performed with a multi-shell diffusion-weighted (DWI) sequence.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera Universitaria Sant'Andrea, Roma

REFERENCES:
- [Background] Dangond F, Donnelly A, Hohlfeld R, Lubetzki C, Kohlhaas S, Leocani L, Ciccarelli O, Stankoff B, Sormani MP, Chataway J, Bozzoli F, Cucca F, Melton L, Coetzee T, Salvetti M. Facing the urgency of therapies for progressive MS - a Progressive MS Alliance proposal. Nat Rev Neurol. 2021 Mar;17(3):185-192. doi: 10.1038/s41582-020-00446-9. Epub 2021 Jan 22. PMID 33483719
- [Background] University of California, San Francisco MS-EPIC Team; Cree BAC, Hollenbach JA, Bove R, Kirkish G, Sacco S, Caverzasi E, Bischof A, Gundel T, Zhu AH, Papinutto N, Stern WA, Bevan C, Romeo A, Goodin DS, Gelfand JM, Graves J, Green AJ, Wilson MR, Zamvil SS, Zhao C, Gomez R, Ragan NR, Rush GQ, Barba P, Santaniello A, Baranzini SE, Oksenberg JR, Henry RG, Hauser SL. Silent progression in disease activity-free relapsing multiple sclerosis. Ann Neurol. 2019 May;85(5):653-666. doi: 10.1002/ana.25463. Epub 2019 Mar 30. PMID 30851128
- [Background] Kappos L, Wolinsky JS, Giovannoni G, Arnold DL, Wang Q, Bernasconi C, Model F, Koendgen H, Manfrini M, Belachew S, Hauser SL. Contribution of Relapse-Independent Progression vs Relapse-Associated Worsening to Overall Confirmed Disability Accumulation in Typical Relapsing Multiple Sclerosis in a Pooled Analysis of 2 Randomized Clinical Trials. JAMA Neurol. 2020 Sep 1;77(9):1132-1140. doi: 10.1001/jamaneurol.2020.1568. PMID 32511687
- [Background] Green AJ. Potential Benefits of Early Aggressive Treatment in Multiple Sclerosis. JAMA Neurol. 2019 Mar 1;76(3):254-256. doi: 10.1001/jamaneurol.2018.4932. No abstract available. PMID 30644966
- [Background] Singh NK, Bracker CA, Hasegawa PM, Handa AK, Buckel S, Hermodson MA, Pfankoch E, Regnier FE, Bressan RA. Characterization of osmotin : a thaumatin-like protein associated with osmotic adaptation in plant cells. Plant Physiol. 1987 Oct;85(2):529-36. doi: 10.1104/pp.85.2.529. PMID 16665731
- [Background] Narasimhan ML, Coca MA, Jin J, Yamauchi T, Ito Y, Kadowaki T, Kim KK, Pardo JM, Damsz B, Hasegawa PM, Yun DJ, Bressan RA. Osmotin is a homolog of mammalian adiponectin and controls apoptosis in yeast through a homolog of mammalian adiponectin receptor. Mol Cell. 2005 Jan 21;17(2):171-80. doi: 10.1016/j.molcel.2004.11.050. PMID 15664187
- [Background] Carbone F, La Rocca C, Matarese G. Immunological functions of leptin and adiponectin. Biochimie. 2012 Oct;94(10):2082-8. doi: 10.1016/j.biochi.2012.05.018. Epub 2012 Jun 26. PMID 22750129
- [Background] Takahashi Y, Watanabe R, Sato Y, Ozawa N, Kojima M, Watanabe-Kominato K, Shirai R, Sato K, Hirano T, Watanabe T. Novel phytopeptide osmotin mimics preventive effects of adiponectin on vascular inflammation and atherosclerosis. Metabolism. 2018 Jun;83:128-138. doi: 10.1016/j.metabol.2018.01.010. Epub 2018 Feb 2. PMID 29410350
- [Background] Liu J, Sui H, Zhao J, Wang Y. Osmotin Protects H9c2 Cells from Simulated Ischemia-Reperfusion Injury through AdipoR1/PI3K/AKT Signaling Pathway. Front Physiol. 2017 Sep 25;8:611. doi: 10.3389/fphys.2017.00611. eCollection 2017. PMID 28993734
- [Background] Badshah H, Ali T, Kim MO. Osmotin attenuates LPS-induced neuroinflammation and memory impairments via the TLR4/NFkappaB signaling pathway. Sci Rep. 2016 Apr 20;6:24493. doi: 10.1038/srep24493. PMID 27093924
- [Background] Fantuzzi G. Adiponectin and inflammation: consensus and controversy. J Allergy Clin Immunol. 2008 Feb;121(2):326-30. doi: 10.1016/j.jaci.2007.10.018. Epub 2007 Dec 3. PMID 18061654
- [Background] Neumeier M, Weigert J, Schaffler A, Wehrwein G, Muller-Ladner U, Scholmerich J, Wrede C, Buechler C. Different effects of adiponectin isoforms in human monocytic cells. J Leukoc Biol. 2006 Apr;79(4):803-8. doi: 10.1189/jlb.0905521. Epub 2006 Jan 24. PMID 16434692
- [Background] Song H, Chan J, Rovin BH. Induction of chemokine expression by adiponectin in vitro is isoform dependent. Transl Res. 2009 Jul;154(1):18-26. doi: 10.1016/j.trsl.2009.04.003. Epub 2009 May 9. PMID 19524870
- [Background] Piccio L, Stark JL, Cross AH. Chronic calorie restriction attenuates experimental autoimmune encephalomyelitis. J Leukoc Biol. 2008 Oct;84(4):940-8. doi: 10.1189/jlb.0208133. Epub 2008 Aug 4. PMID 18678605
- [Background] Hietaharju A, Kuusisto H, Nieminen R, Vuolteenaho K, Elovaara I, Moilanen E. Elevated cerebrospinal fluid adiponectin and adipsin levels in patients with multiple sclerosis: a Finnish co-twin study. Eur J Neurol. 2010 Feb;17(2):332-4. doi: 10.1111/j.1468-1331.2009.02701.x. Epub 2009 Jun 15. PMID 19538214
- [Background] Piccio L, Cantoni C, Henderson JG, Hawiger D, Ramsbottom M, Mikesell R, Ryu J, Hsieh CS, Cremasco V, Haynes W, Dong LQ, Chan L, Galimberti D, Cross AH. Lack of adiponectin leads to increased lymphocyte activation and increased disease severity in a mouse model of multiple sclerosis. Eur J Immunol. 2013 Aug;43(8):2089-100. doi: 10.1002/eji.201242836. Epub 2013 Jun 7. PMID 23640763
- [Background] Devorak J, Mokry LE, Morris JA, Forgetta V, Davey Smith G, Sawcer S, Richards JB. Large differences in adiponectin levels have no clear effect on multiple sclerosis risk: A Mendelian randomization study. Mult Scler. 2017 Oct;23(11):1461-1468. doi: 10.1177/1352458516681196. Epub 2016 Dec 7. PMID 27903934
- [Background] Coban A, Duzel B, Tuzun E, Tamam Y. Investigation of the prognostic value of adipokines in multiple sclerosis. Mult Scler Relat Disord. 2017 Jul;15:11-14. doi: 10.1016/j.msard.2017.04.006. Epub 2017 Apr 20. PMID 28641765
- [Background] Kvistad SS, Myhr KM, Holmoy T, Benth JS, Wergeland S, Beiske AG, Bjerve KS, Hovdal H, Midgard R, Sagen JV, Torkildsen O. Serum levels of leptin and adiponectin are not associated with disease activity or treatment response in multiple sclerosis. J Neuroimmunol. 2018 Oct 15;323:73-77. doi: 10.1016/j.jneuroim.2018.07.011. Epub 2018 Jul 24. PMID 30196837
- [Background] Signoriello E, Lus G, Polito R, Casertano S, Scudiero O, Coletta M, Monaco ML, Rossi F, Nigro E, Daniele A. Adiponectin profile at baseline is correlated to progression and severity of multiple sclerosis. Eur J Neurol. 2019 Feb;26(2):348-355. doi: 10.1111/ene.13822. Epub 2018 Nov 27. PMID 30300462
- [Background] Keyhanian K, Saxena S, Gombolay G, Healy BC, Misra M, Chitnis T. Adipokines are associated with pediatric multiple sclerosis risk and course. Mult Scler Relat Disord. 2019 Nov;36:101384. doi: 10.1016/j.msard.2019.101384. Epub 2019 Sep 5. PMID 31550559
- [Background] Signoriello E, Mallardo M, Nigro E, Polito R, Casertano S, Di Pietro A, Coletta M, Monaco ML, Rossi F, Lus G, Daniele A. Adiponectin in Cerebrospinal Fluid from Patients Affected by Multiple Sclerosis Is Correlated with the Progression and Severity of Disease. Mol Neurobiol. 2021 Jun;58(6):2663-2670. doi: 10.1007/s12035-021-02287-z. Epub 2021 Jan 23. PMID 33486671
- [Background] Nyirenda MH, Fadda G, Healy LM, Mexhitaj I, Poliquin-Lasnier L, Hanwell H, Saveriano AW, Rozenberg A, Li R, Moore CS, Belabani C, Johnson T, O'Mahony J, Arnold DL, Yeh EA, Marrie RA, Dunn S, Banwell B, Bar-Or A. Pro-inflammatory adiponectin in pediatric-onset multiple sclerosis. Mult Scler. 2021 Oct;27(12):1948-1959. doi: 10.1177/1352458521989090. Epub 2021 Feb 1. PMID 33522403
- [Background] Kwon KC, Daniell H. Oral Delivery of Protein Drugs Bioencapsulated in Plant Cells. Mol Ther. 2016 Aug;24(8):1342-50. doi: 10.1038/mt.2016.115. Epub 2016 Jun 6. PMID 27378236
- [Background] Harroud A, Manousaki D, Butler-Laporte G, Mitchell RE, Davey Smith G, Richards JB, Baranzini SE. The relative contributions of obesity, vitamin D, leptin, and adiponectin to multiple sclerosis risk: A Mendelian randomization mediation analysis. Mult Scler. 2021 Nov;27(13):1994-2000. doi: 10.1177/1352458521995484. Epub 2021 Feb 19. PMID 33605807
- [Background] Kim HK, Bae MJ, Lim S, Lee W, Kim S. A Water-Soluble Extract from Actinidia arguta Ameliorates Psoriasis-Like Skin Inflammation in Mice by Inhibition of Neutrophil Infiltration. Nutrients. 2018 Oct 2;10(10):1399. doi: 10.3390/nu10101399. PMID 30279326
- [Background] Parida S, Siddharth S, Sharma D. Adiponectin, Obesity, and Cancer: Clash of the Bigwigs in Health and Disease. Int J Mol Sci. 2019 May 22;20(10):2519. doi: 10.3390/ijms20102519. PMID 31121868
- [Background] Miele M, Costantini S, Colonna G. Structural and functional similarities between osmotin from Nicotiana tabacum seeds and human adiponectin. PLoS One. 2011 Feb 2;6(2):e16690. doi: 10.1371/journal.pone.0016690. PMID 21311758
- [Background] Bhattacharya A, Saini U, Joshi R, Kaur D, Pal AK, Kumar N, Gulati A, Mohanpuria P, Yadav SK, Kumar S, Ahuja PS. Osmotin-expressing transgenic tea plants have improved stress tolerance and are of higher quality. Transgenic Res. 2014 Apr;23(2):211-23. doi: 10.1007/s11248-013-9740-5. Epub 2013 Aug 27. PMID 23982743
- [Derived] Costa V, Aluan K, Schiavetti I, Bason C, Vigo T, Leveraro E, Cabona C, Prada V, Costagli M, Boccia VD, Ruggiero B, Brichetto G, Salvetti M, Sormani MP, Mancardi G, Inglese M, Battaglia MA. Study protocol: Exploratory trial of Forza, an osmotin-based nutraceutical as adjuvant for the treatment of progressive multiple sclerosis. PLoS One. 2025 Feb 27;20(2):e0311214. doi: 10.1371/journal.pone.0311214. eCollection 2025. PMID 40014609